CLINICAL TRIAL: NCT02644707
Title: L-selenomethionine Supplementation in Children and Adolescents With Autoimmune Thyroiditis: a Randomized Blind Placebo-controlled Clinical Trial
Brief Title: Selenium Supplementation in Youths With Autoimmune Thyroiditis
Acronym: THYROSEL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Assimina Galli-Tsinopoulou, ASSSOCIATE PROFESSOR, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARISTOTLE UNIVERSITY
Record Dates: First submitted 2015-12-29; First posted 2016-01-01 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Autoimmune Thyroiditis
MeSH Terms: conditions — Thyroiditis, Autoimmune | interventions — Selenium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- L-selenomethionine (Experimental): A group randomized to receive organic selenium in the form of L-selenomethionine at the dose of 200mcg daily (intervention group) for 6 months
  Interventions: Dietary Supplement: L-selenomethionine
- Placebo (Placebo Comparator): A group randomized to receive placebo (control group) for 6 months
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: L-selenomethionine — The group will be randomized to receive organic selenium in the form of L-selenomethionine at the dose of 200mcg daily (intervention group) for 6 months
  Arms: L-selenomethionine
Other: Placebo — The group will be randomized to receive placebo (control group) for 6 months
  Arms: Placebo

SUMMARY:
To investigate whether the supplementation of organic selenium at the "adult" dose (200 mcg per day in the form of L-selenomethionine) has a favorable impact on thyroid function, including the titer of anti-thyroid antibodies [Anti-thyroid peroxidase (anti-TPO) and Anti-thyroglobulin (anti-Tg) antibodies], in children and adolescents with autoimmune thyroiditis (AT).

DETAILED DESCRIPTION:
Background: Selenium in the form of seleno-cysteine is an essential component of enzymes that remove toxic substances from the body, such as glutathione peroxidase (GPX) in thyroid cells as well as seleno-dependent iodothyronine deiodinase that catalyses extra-thyroidal production of triiodothyronine (T3). In general, selenium deficiency may influence production of free radicals, conversion of thyroxine T4 to T3, cytokine production and immune mechanisms. Thus, it has been previously suggested that its supplementation may have a beneficial effect in patients with autoimmune thyroiditis, especially in those with increased inflammatory activity and a higher antibody titer. Although the two studies that have so far been conducted in pediatric populations demonstrated no significant effect of selenium administration on the titre of antibodies, the researchers did administer selenium either in the form of inorganic sodium selenite at the "adult" dose (100-200 mcg daily) or in the form of organic L-selenomethionine at the reduced dose (50 mcg daily). Therefore, to the best of our knowledge, selenium supplementation in the form of organic L-selenomethionine at the "adult" dose (200 mcg daily) has not been investigated in children and adolescents with autoimmune thyroiditis (AT) so far.

Objective: Our aim is to investigate whether the supplementation of organic selenium at the "adult" dose (200 mcg per day in the form of L-selenomethionine) has a favorable impact on thyroid function, including the titer of anti-thyroid antibodies (thyroid-peroxidase antiTPO, and thyroglobulin -antiTg- antibodies), in children and adolescents with autoimmune thyroiditis (AT).

Design and Methods: This is a randomized blinded placebo-controlled clinical trial of selenium supplementation versus placebo in children and adolescents with autoimmune thyroiditis (AT). The trial will include 100 consecutive participants (50 participants in each arm) from the Unit of Pediatric Endocrinology of the 4th Department of Pediatrics, Medical School, Aristotle University of Thessaloniki, Greece. The patients will be informed and given their written consent to be included in the study. The subjects will then be randomized to receive either organic selenium in the form of L-selenomethionine at the dose of 200mcg daily (intervention group) or placebo (control group) for 6 months. Both groups will receive oral tablets (one daily), which will be identical in appearance, taste and smell and will differ only in the type of active substance (L-selenomethionine or placebo). Six months of additional follow-up will lead to trial duration of 12 months. The experimental supplement will be given by the Pharmaceutical company marketing the product SEMED200® (INTERMED Pharmaceutical Laboratories). In all participants, determination of the concentrations of thyroid-stimulating hormone (TSH), free thyroxine (fT4), thyroid peroxidase antibodies (TPOAb), thyroglobulin antibody (TgAb) will be made at four times (0, 3, 6 and 12 months). Thyroid volume and morphology will also be sonographically evaluated in three times (0, 6 and 12 months). Serum selenium levels in the form of selenomethionine will also be determined once (at the beginning of the study).

Time-schedule: January- February 2015: protocol preparation. March 2015: first participant's first visit. March 2016: last participant's first visit. September 2016: last participant's last visit. September - October 2016: analysis of biological samples and data, preparation of manuscripts, March 2017: last participant's completion of follow-up.

ELIGIBILITY:
Inclusion Criteria: A positive titer of antithyroid peroxidase (anti-TPO) or antithyroglobulin (anti-Tg) antibodies (TPO and / or Tg> 60 IU / ml) and at least one of:

* Abnormal thyroid function that requires substitution treatment with L-thyroxine (TSH > 5 micro-units per milliliter (mcU/ml) and decreased or normal levels of fT4 or fT3)
* Increased volume of thyroid gland (goiter)
* Morphological changes on ultrasound of the thyroid gland

Exclusion Criteria:

* Presence of another chronic disease or autoimmune disease or being under medication
* Age of diagnosis above 18 years

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2014-08; Primary Completion 2016-10 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Change in titer of thyroid autoantibodies (thyroid-peroxidase -AntiTPO-, and thyroglobulin -antiTg- antibodies) | 0,3,6,12 months

SECONDARY OUTCOMES:
Measurement of serum selenium levels | 0 months
Change in state of thyroid function (Euthyroid or Hypothyroid) | 0,6,12 months
  Hypothyroid state will be defined as the state of abnormal thyroid function that requires substitution treatment with L-thyroxine; in particular, if thyroid-stimulating hormone (TSH) serum levels are greater than 5 micro-units per milliliter (mcU/ml) and/or the levels of fT4 or fT3 are decreased. Otherwise the state will be considered as euthyroid.
Change in thyroxine dose per kg per day | 0,6,12 months
Change in thyroid volume measured by ultrasonography | 0,6,12 months

CONTACTS AND LOCATIONS:
Overall Officials: Assimina Galli-Tsinopoulou, Assoc Prof, Principal Investigator — Unit of Pediatric Endocrinology, Diabetes and Metabolism - 4th Department of Pediatrics, Medical School of Aristotle University of Thessaloniki, 56403 Thessaloniki, Greece
Locations (1):
- Unit of Pediatric Endocrinology, Diabetes and Metabolism-4th Department of Pediatrics, Medical School of Aristotle University of Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karanikas G, Schuetz M, Kontur S, Duan H, Kommata S, Schoen R, Antoni A, Kletter K, Dudczak R, Willheim M. No immunological benefit of selenium in consecutive patients with autoimmune thyroiditis. Thyroid. 2008 Jan;18(1):7-12. doi: 10.1089/thy.2007.0127. PMID 18302514
- [Result] Anastasilakis AD, Toulis KA, Nisianakis P, Goulis DG, Kampas L, Valeri RM, Oikonomou D, Tzellos TG, Delaroudis S. Selenomethionine treatment in patients with autoimmune thyroiditis: a prospective, quasi-randomised trial. Int J Clin Pract. 2012 Apr;66(4):378-83. doi: 10.1111/j.1742-1241.2011.02879.x. Epub 2012 Feb 22. PMID 22356267
- [Result] Bonfig W, Gartner R, Schmidt H. Selenium supplementation does not decrease thyroid peroxidase antibody concentration in children and adolescents with autoimmune thyroiditis. ScientificWorldJournal. 2010 Jun 1;10:990-6. doi: 10.1100/tsw.2010.91. PMID 20526530
- [Result] Duntas LH, Mantzou E, Koutras DA. Effects of a six month treatment with selenomethionine in patients with autoimmune thyroiditis. Eur J Endocrinol. 2003 Apr;148(4):389-93. doi: 10.1530/eje.0.1480389. PMID 12656658
- [Result] Eskes SA, Endert E, Fliers E, Birnie E, Hollenbach B, Schomburg L, Kohrle J, Wiersinga WM. Selenite supplementation in euthyroid subjects with thyroid peroxidase antibodies. Clin Endocrinol (Oxf). 2014 Mar;80(3):444-51. doi: 10.1111/cen.12284. Epub 2013 Jul 31. PMID 23844613
- [Result] Gartner R, Gasnier BC, Dietrich JW, Krebs B, Angstwurm MW. Selenium supplementation in patients with autoimmune thyroiditis decreases thyroid peroxidase antibodies concentrations. J Clin Endocrinol Metab. 2002 Apr;87(4):1687-91. doi: 10.1210/jcem.87.4.8421. PMID 11932302
- [Result] Krysiak R, Okopien B. The effect of levothyroxine and selenomethionine on lymphocyte and monocyte cytokine release in women with Hashimoto's thyroiditis. J Clin Endocrinol Metab. 2011 Jul;96(7):2206-15. doi: 10.1210/jc.2010-2986. Epub 2011 Apr 20. PMID 21508145
- [Result] Mazokopakis EE, Papadakis JA, Papadomanolaki MG, Batistakis AG, Giannakopoulos TG, Protopapadakis EE, Ganotakis ES. Effects of 12 months treatment with L-selenomethionine on serum anti-TPO Levels in Patients with Hashimoto's thyroiditis. Thyroid. 2007 Jul;17(7):609-12. doi: 10.1089/thy.2007.0040. PMID 17696828
- [Result] Nacamulli D, Mian C, Petricca D, Lazzarotto F, Barollo S, Pozza D, Masiero S, Faggian D, Plebani M, Girelli ME, Mantero F, Betterle C. Influence of physiological dietary selenium supplementation on the natural course of autoimmune thyroiditis. Clin Endocrinol (Oxf). 2010 Oct;73(4):535-9. doi: 10.1111/j.1365-2265.2009.03758.x. PMID 20039895
- [Result] Negro R, Greco G, Mangieri T, Pezzarossa A, Dazzi D, Hassan H. The influence of selenium supplementation on postpartum thyroid status in pregnant women with thyroid peroxidase autoantibodies. J Clin Endocrinol Metab. 2007 Apr;92(4):1263-8. doi: 10.1210/jc.2006-1821. Epub 2007 Feb 6. PMID 17284630
- [Result] Onal H, Keskindemirci G, Adal E, Ersen A, Korkmaz O. Effects of selenium supplementation in the early stage of autoimmune thyroiditis in childhood: an open-label pilot study. J Pediatr Endocrinol Metab. 2012;25(7-8):639-44. doi: 10.1515/jpem-2012-0078. PMID 23155687
- [Result] Toulis KA, Anastasilakis AD, Tzellos TG, Goulis DG, Kouvelas D. Selenium supplementation in the treatment of Hashimoto's thyroiditis: a systematic review and a meta-analysis. Thyroid. 2010 Oct;20(10):1163-73. doi: 10.1089/thy.2009.0351. PMID 20883174
- [Result] Turker O, Kumanlioglu K, Karapolat I, Dogan I. Selenium treatment in autoimmune thyroiditis: 9-month follow-up with variable doses. J Endocrinol. 2006 Jul;190(1):151-6. doi: 10.1677/joe.1.06661. PMID 16837619
- [Result] van Zuuren EJ, Albusta AY, Fedorowicz Z, Carter B, Pijl H. Selenium supplementation for Hashimoto's thyroiditis. Cochrane Database Syst Rev. 2013 Jun 6;2013(6):CD010223. doi: 10.1002/14651858.CD010223.pub2. PMID 23744563
- [Result] Zhu L, Bai X, Teng WP, Shan ZY, Wang WW, Fan CL, Wang H, Zhang HM. [Effects of selenium supplementation on antibodies of autoimmune thyroiditis]. Zhonghua Yi Xue Za Zhi. 2012 Aug 28;92(32):2256-60. Chinese. PMID 23158484